CLINICAL TRIAL: NCT05076097
Title: A Prospective Phase II Clinical Study of Orelabrutinib in Combination With Lenalidomide and Rituximab (OLR) in First-line Treatment of Mantle Cell Lymphoma
Brief Title: A Study of OLR in First-line Treatment of Mantle Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TS024
Record Dates: First submitted 2021-09-30; First posted 2021-10-13 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-09

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — orelabrutinib; Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orelabtutinib in combination of rituximab and lenalidomide(OLR) Arm (Experimental): Induction phase of mantle cell L lymphoma: Orelabrutinib: 150mg QD D1-28; Lenalidomide: Cycle 1: 15mg QD D1-21, if no dose-limiting toxicity occurred in Cycle 1, cycle 2-6: 20mg QD D1-21; Cycle 1: 375 mg/m2 d1, 8,15,22; Cycle 3, 5: 375 mg/m2 D1 Maintenance treatment phase: Orelabrutinib: 150mg QD D1-28; Lenalidomide: cycle 7-24: 15mg QD D1-21; Cycle 7, 9, 11, 13, 15, 17, 19, 21, 23: 375 mg/m2 D1
  Interventions: Drug: Orelabrutinib in in combination of rituximab and lenalidomide(OLR)

INTERVENTIONS:
Drug: Orelabrutinib in in combination of rituximab and lenalidomide(OLR) — Induction treatment phase: Orelabrutinib: 150mg QD D1-28; Lenalidomide: Cycle 1: 15mg QD D1-21, if no dose-limiting toxicity occurred in Cycle 1, cycle 2-6: 20mg QD D1-21; Cycle 1: 375 mg/m2 d1, 8,15,22; Cycle 3, 5: 375 mg/m2 D1 Maintenance treatment phase: Orelabrutinib: 150mg QD D1-28; Lenalidomide: cycle 7-24: 15mg QD D1-21; Cycle 7, 9, 11, 13, 15, 17, 19, 21, 23: 375 mg/m2 D1. 28 days for a cycle.
  Other Names: OLR Arm

SUMMARY:
This is a single-arm, multicenter, open label phase II clinical study to evaluate the efficacy and safety of OLR in the treatment of initially treated mantle cell lymphoma.

DETAILED DESCRIPTION:
Patients initially treated with mantle cell lymphoma were screened for OLR regimen according to study admission criteria. The study will accept up to 24 cycles of treatment until disease progression or intolerable toxicity occurs and subjects voluntarily withdraw informed consent. Patients undergoing hematopoietic stem cell transplantation after complete remission may begin stem cell collection after induction therapy for at least 6 months. Twenty-nine patients are expected to be enrolled

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed mantle cell lymphoma with chromosomal translocation. All subjects must provide adequate archived or fresh tumor tissue samples for immunohistochemistry (IHC) testing.
2. Age 18-70, both male and female.
3. No previous systemic treatment for lymphoma.
4. Have at least one measurable lesion. Measurable disease was defined as measurable tumor masses ≥1.5 cm in one or both dimensions and measurable spleen lesions.
5. Eastern Oncology Collaboration group physical status score was 0-2.
6. Adequate hematological function
7. Life expectancy >3 months.
8. Have the ability to provide written informed consent and understand and comply with study requirements.
9. Ability to adhere to research visit schedules and other protocol requirements

Exclusion Criteria:

1. Histology conformed blastolytic mantle cell lymphoma and polymorphic mantle cell lymphoma.
2. Patients with current or suspected central nervous system involvement and history of this disease
3. Received Bruton's tyrosine kinase inhibitor treatment
4. Receive lenalidomide treatment
5. Received other anti-tumor treatments
6. Major surgery within 4 weeks prior to screening.
7. Have a history of other active malignant diseases within 2 years prior to study entry,
8. Systemic fungal, bacterial or viral infection with uncontrolled activity
9. The following serological states are known for human immunodeficiency virus (HIV) infection or suggest the presence of active hepatitis B or C virus infection
10. Clinically serious cardiovascular disease
11. A history of severe hemorrhagic disorders, such as hemophilia A, hemophilia B, von willebrand disease, or A history of spontaneous bleeding requiring blood transfusion or other medical intervention.
12. A history of deep vein thrombosis (DVT) or pulmonary embolism (PE) within the past 12 months.
13. A history of major cerebrovascular disease/event, including stroke or intracranial hemorrhage, in the 6 months prior to first administration of the study drug.
14. Anticoagulant therapy with warfarin or an equivalent vitamin K antagonist or anticoagulant therapy is required within 7 days of initial use of the study drug.
15. Pregnant or lactating women
16. Hypersensitivity to any study drug
17. The presence of any life-threatening disease, medical condition, or organ system dysfunction that the investigator considers to be likely to affect the safety of the subject or cause risk

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-10-15 (Estimated); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
Complete Response Rate | At the end of Cycle 6(each cycle is 28 days)
  The proportion of patients receiving the treatment with complete remission

SECONDARY OUTCOMES:
Objective Response Rate | Approximately 2 years
  The proportion of patients with response of PR and CR.
Time to Response | Approximately 1 year
  Measured from the date of initiation of treatment to the time of response
The Progression Free Survival Rate in 2 Years | 2 Years
  The proportion of patients who didn't achieve disease progression or death in 2 years.
The Overall Survival Rate in 2 Years | 2 Years
  The proportion of patients who didn't achieve death in 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Huilai Zhang, PHD, Principal Investigator — Director of Hematology Department
Locations (1):
- Tianjin Medical University Cancer Insititute & Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No
No individual patient data will be shared with other researchers

REFERENCES:
- [Background] 2020 ASH, poster 2042
- [Background] EHA 2020-Abstract S228
- [Result] Al-Hamadani M, Habermann TM, Cerhan JR, Macon WR, Maurer MJ, Go RS. Non-Hodgkin lymphoma subtype distribution, geodemographic patterns, and survival in the US: A longitudinal analysis of the National Cancer Data Base from 1998 to 2011. Am J Hematol. 2015 Sep;90(9):790-5. doi: 10.1002/ajh.24086. Epub 2015 Jul 27. PMID 26096944